CLINICAL TRIAL: NCT00201812
Title: Phase I & Biological Study of Etanercept & Weekly Docetaxel in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0023
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Tumors
Keywords: Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — Etanercept; Docetaxel; Dexamethasone; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Etanercept — 7 days prior to treatment with docetaxel. Administered twice weekly throughout the study.
  Other Names: Enbrel
Drug: Docetaxel — Administered intervenously (IV) over 30 minutes through an infusion pump once a week (every 7 days). A cycle will comprise six weekly treatments followed by 2 weeks of rest.
  Other Names: Taxotere
Drug: Dexamethasone — Administered orally 8 mg 12 hours prior to docetaxel, immediately prior to docetaxel (two hours after etanercept), and 12 hours after docetaxel to complete a total of 3 doses (total dose 24 mg/week) on treatment weeks.
  Other Names: steriod; glucocorticoid

SUMMARY:
To determine the safety and efficacy of the combination of Etanercept and Docetaxel in patients with advanced solid tumors for which there is no standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have pathologically or cytologically confirmed advanced solid malignancy for which there is no standard treatment exists.
* Solid malignancy that has persisted or recurred following prior therapy or advanced solid malignancy for which docetaxel is considered an acceptable first line treatment option:

  * Non-Small Cell Lung
  * Breast
  * Head and Neck
  * Esophageal
  * Stomach
  * Ovarian carcinomas
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Life expectancy of at least 12 weeks.
* Must have adequate organ function
* Peripheral Neuropathy must be less than Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-11; Primary Completion 2004-01 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD) of weekly docetaxel in combination with etanercept. | up to 4 years

SECONDARY OUTCOMES:
Characterize toxicities of weekly docetaxel when administered weekly to patients with solid malignancies to determine if co-administration of etanercept can result in higher tolerated doses of docetaxel. | up to 4 years
Determine if weekly docetaxel administration is associated with increased expression of TNF and if inactivation of TNF by etanercept is associated with a decrease in the rate of moderate to severe asthenia. | up to 4 years
Preliminarily evaluate antitumor activity for docetaxel in combination with etanercept. | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Villalona, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Monk JP, Phillips G, Waite R, Kuhn J, Schaaf LJ, Otterson GA, Guttridge D, Rhoades C, Shah M, Criswell T, Caligiuri MA, Villalona-Calero MA. Assessment of tumor necrosis factor alpha blockade as an intervention to improve tolerability of dose-intensive chemotherapy in cancer patients. J Clin Oncol. 2006 Apr 20;24(12):1852-9. doi: 10.1200/JCO.2005.04.2838. PMID 16622259
- See also: Jamesline — http://cancer.osu.edu